CLINICAL TRIAL: NCT06712524
Title: A Prospective Real-world Study of the Effect of Different Surgical Approaches on the Recurrence Rate and Aesthetic Outcome of Granulomatous Mastitis
Brief Title: Effect of Different Surgical Approaches of Granulomatous Mastitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hongmei Zheng, PhD, Doctor, Hubei Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLHBCH2024YN-093
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Breast-conserving Plastic Surgery; Granulomatous Mastitis
Keywords: Granulomatous mastitis; breast conserving plastic surgery; Aesthetics scores
MeSH Terms: conditions — Granulomatous Mastitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast-conserving plastic surgery group (Experimental): Breast-conserving plastic surgery
  Interventions: Procedure: Breast-conserving plastic surgery
- Traditional breast surgery group (Active Comparator): Traditional breast surgery
  Interventions: Procedure: Traditional breast surgery

INTERVENTIONS:
Procedure: Breast-conserving plastic surgery — The commonly used breast conserving plastic surgery includes tennis racket, bat wing, V/J breast plasty, Grisotti and so on.
  Arms: Breast-conserving plastic surgery group
Procedure: Traditional breast surgery — Traditional breast surgery
  Arms: Traditional breast surgery group

SUMMARY:
The objective of this study was to prospectively investigate the effects of different surgical approaches on the recurrence rate and aesthetic outcome of patients with granulomatous mastitis. The patients were divided into traditional surgery group and plastic surgery group.

DETAILED DESCRIPTION:
Granulomatous mastitis is a rare benign inflammatory breast disease first described by Kessler and Wollock in 1972. It resembles inflammatory breast cancer disease in imaging and mainly affects women of childbearing age. Treatment methods include steroid therapy, antibiotics and surgical treatment. However, due to the adverse reactions of drug treatment and the high recurrence rate after traditional surgery, there is no definitive preferred treatment form at present, and most clinicians are still in the stage of empirical treatment.

Breast-conserving plastic surgery has been widely used by surgeons because it can remove a larger range of breast cancer, so it has higher safety and aesthetics compared with traditional breast conserving surgery. So, if patients with mastitis are treated surgically, will they also benefit from breast-conserving surgery? At present, the commonly used breast conserving plastic surgery includes tennis racket, bat wing, V/J breast plasty, Grisotti and so on. Therefore, this study prospectively grouped mastitis patients who selected surgery, and divided them into traditional surgery group and plastic breast-conserving surgery group. The postoperative recurrence, adverse reactions, aesthetics and satisfaction of the two groups were compared.

It is hoped that this study will bring a new research direction for the surgical treatment of mastitis and provide a clearer guiding significance for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

Only the subjects who meet all the following criteria may be included in this study:

1. Ability to understand the study procedures and contents, and willingness to voluntarily sign the written informed consent form;
2. 18≤Age≤75 years old, female;
3. Histologically confirmed granulomatous mastitis;
4. low and moderate risk for anesthesia.

Exclusion Criteria:

The subjects who meet any of the following criteria shall not be included in this study:

1. Absolute and relative contraindication for surgery;
2. Previous history of breast cancer or other malignancies;
3. Pregnancy;
4. Any serious complications which caused patients not suitable to participate this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2, 3, 5 year
  The recurrence rate of mastitis patients was compared between traditional surgery group and plastic surgery group.

SECONDARY OUTCOMES:
Aesthetics scores | 2, 3, 5 year
  The patients' satisfaction and quality of life after surgery were evaluated by BREAST Q questionnaire. The full score is 100, with higher scores indicating higher patient satisfaction and quality of life.
  Occurring rate of complications including the occurring rate of infection, hemorrhage, time in hospital in each group were recorded in patients' medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhong Wu, Doctor, Study Chair — Hubei Cancer Hospital
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Patient information was protected according to the privacy requirements of our unit.